CLINICAL TRIAL: NCT01790698
Title: Improving Outcome of Necrotizing Fasciitis: Elucidation of Complex Host and Pathogen Signatures That Dictate Severity of Tissue Infection
Brief Title: Systems Medicine to Study Necrotizing Soft Tissue Infections (NSTIs).
Acronym: INFECT
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Rigshospitalet, Denmark (Other); Karolinska University Hospital (Other); Blekinge County Council Hospital (Other); Sahlgrenska University Hospital (Other); University of Bergen (Other); Helmholtz Centre for Infection Research (Other); Wageningen University (Other); University of Lyon (Other); LifeGlimmer GmbH (Unknown); Anagnostics Bioanalysis GmbH (Unknown); Lee Spark NF Foundation (Unknown); Tel Aviv University (Other)
Responsible Party: Principal Investigator, Anna Norrby-Teglund, Professor, Coordinator of INFECT, Karolinska Institutet
Other Study IDs: INFECT-FP7305340
Record Dates: First submitted 2013-02-04; First posted 2013-02-13 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Soft Tissue Infections; Necrotizing Fasciitis; Necrotizing Soft Tissue Infections
Keywords: Necrotizing fasciitis; Streptococcus pyogenes; Staphylococcus aureus; Immunopathogenesis
MeSH Terms: conditions — Soft Tissue Infections; Fasciitis, Necrotizing; Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Bacterial isolates, whole blood, plasma, tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
This proposal focuses on highly lethal destructive tissue infections, i.e. necrotizing fasciitis and other necrotizing soft tissue infections (NSTIs), which are associated with high morbidity and mortality. The fulminant course of NSTIs demands immediate diagnosis and adequate interventions in order to salvage lives and limbs. However, diagnosis and management are difficult due to heterogeneity in clinical presentation, in co-morbidities and in microbiological aetiology. Thus, there is an urgent need for novel diagnostics and therapeutics in order to improve outcome of NSTIs. A comprehensive knowledge of diagnostic features, causative microbial agent, treatment strategies, and pathogenic mechanisms (host and bacterial disease traits and their underlying interaction network) is required for an improved diagnosis and management of NSTIs. The current proposal is designed to obtain such insights through an integrated systems biology approach in patients and experimental models. The project is based on a prospective NSTI patients cohort including a clinical registry to document clinical data and treatment strategies, combined with an isolate and biobank collection. The samples will be analyzed through advanced bioinformatics and computational modelling work flow to identify and quantify pathogen signatures and underlying networks that contribute to disease outcome. One aim is to translate clinical and systems biology data into development of novel diagnostics.

DETAILED DESCRIPTION:
Patients will be prospectively recruited at 5 clinical centers (Rigshospitalet, Karolinska University Hospital, Blekinge University, Sahlgrenska University and University of Bergen). Clinical definition criteria for NSTI: NSTI is a clinical diagnosis. Initial signs are the occurrence of erythema, pain or tenderness beyond margins of erythema and swelling. Imaging and laboratory tests have little predictive value in the early stage. The gold standard modality for diagnosis of NSTI remains operative exploration. Operative findings that are consistent with NSTI include "dishwater or foul smelling discharge, necrosis or lack of bleeding and loss of the normal resistance of the fascia to finger dissection. A patient admitted for critical care and / or surgery due to severe soft tissue infection of the fascia, muscle or subcutaneous tissues will be enrolled in this NSTI study. The patients will be stratified based on several clinical parameters including among others SAPS score, presence of multiorgan failure, and hypotensive shock. This stratification serves to classify the patients in defined severity classes to be used in analyses and modeling. Detailed demographic and clinical information will be documented in the interactive database including: age, gender, medical history, clinical presentation (shock, multiorgan failure etc), treatment and outcome. Disease progress: The clinical database is to contain information on the spread of the infection at the different times of inspection/surgical intervention. Severity of the infections will be documented by use of the updated CREST classification scheme, SAPS III score, and the LRINEC score. Detailed information regarding antimicrobial therapy, surgical intervention, innovative therapy (IVIG and HBO) will be documented.

Samples will be collected from all enrolled patients. Standard operating procedures will be generated and implemented at all sites to ensure a quality assured collection and handling of samples. Samples to be collected include (a) isolates, (b) blood samples to be processed for DNA, RNA and plasma/cells and (c) tissue biopsies in all patients whenever surgical interventions are indicated. The samples will be analyzed using genomics, transcriptomics, metabolomics and proteomics.

ELIGIBILITY:
Inclusion Criteria:

Necrotizing soft tissue infections

Exclusion Criteria:

Patients under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with NSTI
Sampling Method: Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2013-01; Primary Completion 2017-06 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Prognostic/diagnostic value (ROC curves: specificity, sensitivity, predictive values) of classification and severity scores in NSTIs | 3 months - further oservation up to 24 month may apply

SECONDARY OUTCOMES:
Effect of IVIG and HBO-therapy on mortality rates in matched (defined by severity scores and aetiology) NSTI patients | 3 months - further observation up to 24 month may apply
Presence of hypotension, multiorgan failure, or fatal outcome of NSTI in relation to microbiologic aetiology | 3 months - further observation up to 60 month may apply

CONTACTS AND LOCATIONS:
Locations (5):
- Rigshospitalet, Copenhagen, Denmark
- University of Bergen, Bergen, Norway
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Blekinge Hospital, Karlskrona
  - Karolinska University Hospital, Stockholm

REFERENCES:
- [Derived] Hyldegaard O, Nekludov M, Arnell P, Nedrebo T, Karlsson Y, Madsen MB, Skrede S, Dos Santos VM, Svensson M, Perner A, Vinkel J, Kjellberg A, Rosen A, Douglas J, Bruun T, Hardt C, Norrby-Teglund A, Hedetoft M. Use of Hyperbaric Oxygen in Patients with Necrotizing Soft Tissue Infections: A Scandinavian Multicenter, Prospective, Observational Cohort. Infect Dis Ther. 2025 Aug;14(8):1715-1738. doi: 10.1007/s40121-025-01184-5. Epub 2025 Jul 4. PMID 40613866
- [Derived] Vinkel J, Buil A, Hyldegaard O. Blood from septic patients with necrotising soft tissue infection treated with hyperbaric oxygen reveal different gene expression patterns compared to standard treatment. BMC Med Genomics. 2025 Jan 14;18(1):12. doi: 10.1186/s12920-024-02075-3. PMID 39810178
- [Derived] Vinkel J, Rib L, Buil A, Hedetoft M, Hyldegaard O. Key pathways and genes that are altered during treatment with hyperbaric oxygen in patients with sepsis due to necrotizing soft tissue infection (HBOmic study). Eur J Med Res. 2023 Nov 10;28(1):507. doi: 10.1186/s40001-023-01466-z. PMID 37946314
- [Derived] Vinkel J, Rib L, Buil A, Hedetoft M, Hyldegaard O. Investigating the Effects of Hyperbaric Oxygen Treatment in Necrotizing Soft Tissue Infection With Transcriptomics and Machine Learning (the HBOmic Study): Protocol for a Prospective Cohort Study With Data Validation. JMIR Res Protoc. 2022 Nov 25;11(11):e39252. doi: 10.2196/39252. PMID 36427229
- [Derived] Palma Medina LM, Rath E, Jahagirdar S, Bruun T, Madsen MB, Stralin K, Unge C, Hansen MB, Arnell P, Nekludov M, Hyldegaard O, Lourda M, Santos VAMD, Saccenti E, Skrede S, Svensson M, Norrby-Teglund A. Discriminatory plasma biomarkers predict specific clinical phenotypes of necrotizing soft-tissue infections. J Clin Invest. 2021 Jul 15;131(14):e149523. doi: 10.1172/JCI149523. PMID 34263738
- [Derived] Bergsten H, Madsen MB, Bergey F, Hyldegaard O, Skrede S, Arnell P, Oppegaard O, Itzek A, Perner A, Svensson M, Norrby-Teglund A; INFECT Study Group. Correlation Between Immunoglobulin Dose Administered and Plasma Neutralization of Streptococcal Superantigens in Patients With Necrotizing Soft Tissue Infections. Clin Infect Dis. 2020 Oct 23;71(7):1772-1775. doi: 10.1093/cid/ciaa022. PMID 31916575
- See also: website of INFECT — http://www.fp7infect.eu